CLINICAL TRIAL: NCT00020501
Title: A Phase III Prospective Random Assignment Trial of Regional and Systemic Chemotherapy With or Without Initial Isolated Hepatic Perfusion for Patients With Metastatic Unresectable Colorectal Cancers of the Liver
Brief Title: Chemotherapy With or Without Isolated Hepatic Perfusion With Melphalan in Treating Patients With Colorectal Cancer That Has Spread to the Liver
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 010093; NCI-01-C-0093; CDR0000068562; NCT00011427 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Floxuridine; Fluorouracil; Irinotecan; Leucovorin; Melphalan; Diathermy

INTERVENTIONS:
Drug: FOLFIRI regimen
Drug: floxuridine
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Drug: melphalan
Procedure: hyperthermia treatment

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving them in different ways may kill more tumor cells. It is not yet known which chemotherapy regimen is most effective for colorectal cancer that has spread to the liver.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without isolated hepatic perfusion with melphalan in treating patients who have colorectal cancer that has spread to the liver.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the disease-free and overall survival of patients with unresectable colorectal cancer metastatic to the liver treated with regional and systemic chemotherapy with or without isolated hepatic perfusion with melphalan.
* Compare the response rate and duration of response in patients treated with these regimens.
* Compare the patterns of recurrence (liver vs systemic) in patients treated with these regimens.
* Compare the health-related quality of life (QOL) of patients treated with these regimens.
* Determine whether baseline QOL correlates with length of survival of patients treated with these regimens.

OUTLINE: This is a randomized study. Patients are stratified according to prior chemotherapy for liver metastasis (yes vs no) and percentage of hepatic replacement (less than 25% vs at least 25%). All patients undergo laparotomy to determine final eligibility. Eligible patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo hyperthermic isolated hepatic perfusion with melphalan over 60 minutes. Patients then undergo placement of an intrahepatic pump or port. At 6 weeks post hepatic perfusion, patients receive systemic chemotherapy comprising irinotecan IV over 90 minutes on day 1 followed by fluorouracil IV over 15 minutes and leucovorin calcium (CF) IV over 15 minutes on days 1-3. Patients receive local chemotherapy comprising floxuridine (FUDR) and CF by hepatic arterial infusion (HAI) continuously on days 14-28.
* Arm II: Patients undergo placement of an intrahepatic pump or port at laparotomy. At 7 days post laparotomy, patients receive FUDR and CF by HAI continuously for 14 days. Beginning 2 weeks after completion of HAI, patients receive systemic and local chemotherapy as in arm I.

Treatment with combined systemic and local chemotherapy repeats every 35 days for a maximum of 6 courses. Treatment with local chemotherapy alone repeats every 28 days for a maximum of 6 additional courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, postoperatively, every third course of chemotherapy, every 3 months for 2 years, and then every 6 months thereafter.

Patients are followed every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 168 patients (84 per treatment arm) will be accrued for this study within 54 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic colorectal cancer of the parenchyma of the liver

  * No evidence of extrahepatic disease (limited resectable extrahepatic disease allowed)
* Unresectable liver metastasis, as defined by the following:

  * More than 3 sites of disease
  * Bilobar disease
  * Tumor abutting major vascular or ductal structures
* Measurable disease
* No biopsy-proven cirrhosis or evidence of significant portal hypertension manifested by ascites, esophageal varices, or collateral vessels around organs drained by the portal venous system

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count greater than 100,000/mm^3
* Hematocrit greater than 27.0%
* WBC greater than 3,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL
* PT no greater than 2 seconds over upper limit of normal
* Elevations in transaminases secondary to metastatic disease allowed
* No veno-occlusive disease
* No active chronic hepatitis

  * Hepatitis B or C allowed provided there is no evidence of cirrhosis

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No ischemic cardiac disease
* No prior congestive heart failure with LVEF less than 40%

Pulmonary:

* No chronic obstructive pulmonary disease or other chronic pulmonary disease with pulmonary function test less than 50% of predicted

Other:

* No active infections
* Not pregnant or nursing
* Negative pregnancy test
* Weight greater than 30 kg

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy for disease and recovered

Chemotherapy:

* At least 4 weeks since prior chemotherapy for disease and recovered
* No prior intrahepatic artery infusion therapy with floxuridine

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy for disease and recovered

Surgery:

* Not specified

Other:

* No concurrent immunosuppressive drugs
* No concurrent chronic anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-03; Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Richard Alexander, MD, FACS, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States